CLINICAL TRIAL: NCT05147038
Title: The Impact of Tele-coaching on the Physical Activity Level in Patients With Chronic Respiratory Disease
Brief Title: The Impact of Tele-coaching on the Physical Activity Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palacky University (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Zdenek Svoboda, Tamara Zlamalova, Palacký University Olomouc, the Department of Physiotherapy, Principal Investigator, Ph.D. student, Palacky University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 80/2020
Record Dates: First submitted 2021-11-09; First posted 2021-12-07 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Telemedicine
Keywords: Tele-coaching; Physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study group is divided into the intervention and control group. A randomisation was stratified according to the disease (Idiopathic Pulmonary Fibrosis (IPF) and non-IPF). At first, the participants undergo an initial assessment including a respiratory muscle function and strength testing, physical activity measurement, fatigue, depression status, overall quality of life, disease status, exercise capacity and isometric quadriceps muscle strength testing. Both groups will receive information about the importance of being physically active and the PA recommendations provided by the World Health Organization (leaflet discussed in an education session (one-to-one) of 10-15 minutes). The intervention and control periods are followed by a final assessment (exactly the same as the initial one).
Masking Description: Neither patients nor investigators will be blinded for the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants allocated into the intervention group will be coached for 12 weeks by a tele-coaching mobile App containing tips for PA increase and for number of steps recording (visual feedback for the patient).
  Interventions: Device: Tele-coaching
- Control group (No Intervention): Participants in the control group will receive usual care (including regular visits) together with the educational information.

INTERVENTIONS:
Device: Tele-coaching — The participants are instructed to use a "Fitbit" fitness tracker to record the number of steps. This device is compatible with the "m-PAC" App, which was developed for this specific group of participants (individuals suffering from a chronic lung disease). The participants receive a feedback via the "m-PAC" App every day and they also receive a week report to be albe to adjust their step goal. They are asked to increase or keep their week goal every Sunday after reviewing a weekly report. The participants also receive tips for their PA improvement and they are asked for medication change specification (every Wednesday).
  Arms: Intervention group

SUMMARY:
The study aims to test the benefits of a semi-automated tele-coaching program to coach adult participants with chronic lung disease towards a more active lifestyle.

DETAILED DESCRIPTION:
The level of physical activity (PA) has been shown to be an important predictor for morbidity and mortality in individuals with chronic respiratory diseases, for instance Chronic Obstructive Pulmonary Disease (COPD) or Idiopathic Pulmonary Fibrosis (IPF). Physical inactivity and sedentary behavior is a common feature of patients with chronic respiratory diseases. Pulmonary rehabilitation is known as a beneficial intervention in exercise capacity, disease symptoms and quality of life in respiratory diseases. Despite the overall large benefits on exercise capacity and other variables described above, it does not automatically translate into increases in PA. Recent literature shows that coaching programs specifically aiming to increase PA are more likely to result in PA changes.

Therefore, this study was designed to investigate the impact of 3-month (12 weeks) tele-coaching intervention on PA level of adult participants suffering from a chronic lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Stable patients, older than 18 years of age, with a diagnosis of interstitial lung disease
* Understands and is able to work with a smart phone application (judged by the investigator)
* On stable pharmacotherapy
* Diffusing capacity of the lungs for carbon monoxide (DLCO) ≥30%predicted

Exclusion Criteria:

* On the waiting list for a lung transplantation
* Life expectancy below 3 months
* Respiratory tract infection or an exacerbation or change in maintenance medication within 4 weeks before study enrolment
* Extra pulmonary impairments, unrelated to the underlying lung disease, interfering with physical activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Objective measurement of physical activity | 12 weeks
  Change in weekly mean step count 12 weeks post randomization in the intervention group as compared to the control group.

SECONDARY OUTCOMES:
Physical activity parameters | 12 weeks
  Objectively measured mean daily time in at least moderate intense activity, walking time, movement intensity and activity bout duration.
Spirometry 1 | 12 weeks
  Respiratory muscle function 1 (VC = vital capacity, FVC = forced vital capacity, FEV1 = forced expiratory volume at one second [L]).
Spirometry 2 | 12 weeks
  Respiratory muscle function 2 (PEF = peak expiratory flow [L/min]).
Spirometry 3 | 12 weeks
  Respiratory muscle strength (MIP = maximum inspiratory pressure, MEP = maximum expiratory pressure, P0.1 = airway occlusion pressure [kPa], TTmus = tension time index).
Six minute walk test | 12 weeks
  Functional exercise capacity.
Isometric Quadriceps force | 12 weeks
  Isometric Quadriceps strength measurement.
Questionnaire 1 | 12 weeks
  Health status evaluation: 36-Item Short Form Survey (SF-36). There are 8 scales. Each scale is directly transformed into a 0-100 scale (each question carries equal weight). The lower the score is, the more disability it expresses.
Questionnaire 2 | 12 weeks
  Interstitial lung disease specific health-related quality of life evaluation: The King's Brief Interstitial Lung Disease (KBILD) questionnaire. A15-item validated questionnaire. The total score ranges from 0-100. There are three domain scores: Psychological, Breathlessness and activities and Chest symptoms. The higher score reflects better health-related quality of life.
Questionnaire 3 | 12 weeks
  Anxiety and depression evaluation: Hospital Anxiety and Depression Scale (HADS). There are 14 items. The scoring ranges from 0 to 21. The higher the score, the more severe the anxiety and depression level is.
Questionnaire 4 | 12 weeks
  Fatigue evaluation: Multidimensional Assessment of Fatigue (MAF) Scale. It contains 16 items. Scores range from 1 (no fatigue) to 50 (severe fatigue) and the higher score means worse fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Culture, Palacky University Olomouc, Olomouc, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Breuls S, Zlamalova T, Raisova K, Blondeel A, Wuyts M, Dvoracek M, Zurkova M, Yserbyt J, Janssens W, Wuyts W, Troosters T, Demeyer H. Physical activity coaching in patients with interstitial lung diseases: A randomized controlled trial. Chron Respir Dis. 2024 Jan-Dec;21:14799731241235231. doi: 10.1177/14799731241235231. PMID 38511242